CLINICAL TRIAL: NCT04359615
Title: Efficacy and Safety of Favipiravir Compared to the Base Therapeutic Regiment in Moderate to Severe COVID-19: A Randomized, Controlled, Double-Blind, Clinical Trial
Brief Title: Favipiravir in Hospitalized COVID-19 Patients
Acronym: FIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Sina Naghibi Irvani, MD, MPH, MBA, Senior Researcher., Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Favipiravir in COVID-19
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; Hydroxychloroquine; Chloroquine; Favipiravir; Novel Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: The present study is a randomized, double-blind, placebo-controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental)
  Interventions: Drug: Favipiravir; Drug: Hydroxychloroquine
- Control (Active Comparator)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Favipiravir — This will be drug only used in the intervention arm of our study, designed mainly to assess the additional efficacy and safety of Favipiravir in COVID-19 patients.
  Arms: Favipiravir
Drug: Hydroxychloroquine — This Drug will be used in all arms as mandated by our governmental guidelines.

SUMMARY:
The present study is a randomized, double-blind, controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

DETAILED DESCRIPTION:
Favipiravir, previously known as T-705, is a prodrug of a purine nucleotide, favipiravir ribofuranosyl-5'-triphosphate. The active agent inhibits the RNA polymerase, halting viral replication. Most of favipiravir's preclinical data are derived from its influenza and Ebola activity; however, the agent also demonstrated broad activity against other RNA viruses. In vitro, the 50% effective concentration (EC50) of favipiravir against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) was 61.88 μM/L in Vero E6 cells.

Limited clinical experience has been reported supporting the use of favipiravir for COVID-19. In a prospective, randomized, multicenter study, favipiravir (n = 120) was compared with Arbidol (n = 120) for the treatment of moderate and severe COVID-19 infections. Differences in clinical recovery at day 7 were observed in patients with moderate infections (71.4% favipiravir and 55.9% Arbidol, P = .019). No significant differences were observed in the severe or severe and moderate (combined) arms.73 These data support further investigation with randomized clinical trials (RCTs) of the efficacy of favipiravir for the treatment of COVID-19.

Chloroquine has been a broadly-utilized anti-malaria agent which back in 2006, had been proved to be a powerful wide-spectrum antiviral. Moreover, Chloroquine has the characteristics of anti-inflammatory and immune-modulatory by inhibiting the production of tumor necrosis factor alpha (TNF-α) along with interleukin 6 (IL-6). In the first half of February, a study illustrated puissant inhibition of SARS-CoV-2 by Chloroquine, when taking two 500-mg tablets of it by mouth per day; similar to some clinical studies in China through this outbreak. According to the news briefing of a study, it was indicated that chloroquine phosphate actually outdo the control treatment in inhibition of pneumonia exacerbation, improving lung imaging findings, and curtailing the disease course. Another study evaluated the possible doses of chloroquine (CQ) and hydroxychloroquine (HCQ) to find the optimized dose in treatment of COVID-19. They revealed that while within in-vitro settings Hydroxychloroquine is more potent than chloroquine. As a conclusion, they suggested a 800 mg daily dose of hydroxychloroquine, followed by an overall maintenance dose of 400 mg per day divided in two separate doses, which was three-fold more potent compared to the 500 mg twice daily administration of chloroquine in 5 days. The new study published in 16th March, pointed out that hydroxychloroquine was notably effectual in eradicating SARS-CoV-2 from the nasopharynx. Currently the evidence is quite inconclusive about the effectiveness or comparative effectiveness of either HCQ or CQ. Moreover, CQ has recently become scarce and even unavailable for ordering due to a huge demand for it, all because of a significant interest gained as a potential medicinal alternative for the management of COVID-19. In spite of all, the primary experience in China and France is propitious for the potential role of chloroquine, or alternatively hydroxychloroquine, for managing COVID-19.

The present study is a randomized, double-blind, controlled, clinical trial, with the approval of the ethics committee will be conducted on patients who have a positive test confirming COVID-19 in Shahid Modarres Medical Education Center and Hospital in Tehran. Patients will be randomly assigned to the two arms of the study and after completing the course of treatment and collecting and analyzing the necessary information from each patient, the results of the study will be published both on this site and in the form of an article in a reputable international journal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* COVID-19 Confirmed Cases (Reverse transcription polymerase chain reaction (RT-PCR) Confirmed).
* Tympanic Temperature of ≥37.5 AND at least one of the following: Cough, Sputum production, nasal discharge, myalgia, headache or fatigue) on admission.
* Time of onset of the symptoms should be acute ( Days ≤ 10).
* SpO2 ≤ 93%
* Respiratory Rate ≥ 22

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present.
* Patients with prolonged QT or PR intervals, Second or Third Degree heart block and Arrhythmias.
* Patients using drugs with potential interaction with Favipiravir or Hydroxychloroquine.
* Pregnant or lactating women.
* History of alcohol or drug addiction in the past 5 years.
* Blood Alanine transaminase/aspartate aminotransferase (ALT/AST) levels > 5 times the upper limit of normal on laboratory results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-05-03 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From date of randomization until 14 days later.
  Improvement of two points on a seven-category ordinal scale (recommended by the World Health Organization: Coronavirus disease (COVID-2019) R&D. Geneva: World Health Organization) or discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Mortality | From date of randomization until 14 days later.
  If the patient dies, we have reached an outcome.
oxygen saturation by pulse oximetry (SpO2) Improvement | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  Pulse-oxymetry
Incidence of new mechanical ventilation use | From date of randomization until 14 days later.
  Incidence of new mechanical ventilation use
Duration of hospitalization | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 14 days.
  Duration of hospitalization (days)
Cumulative incidence of serious adverse events | Days 1, 2, 3, 4, 5, 6, 7 and 14.
  With incidence of any serious adverse effects, the outcome has happened.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Fathi, MD, Study Chair — Shahid Beheshti University of Medical Sciences; Sasan Tavana, MD, Study Director — Shahid Beheshti University of Medical Sciences; Nasser Malekpour Alamdari, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mehran Lack, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Nader Markazi, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Sanaz Zargar Balaye Jam, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Seyed Sina Naghibi Irvani, MD, MPH, MBA, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Modarres Hospital, Shahid Beheshti University of Medical Sciences and Health Services, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided
There is no further information.